CLINICAL TRIAL: NCT00005602
Title: Phase I Study of Concurrent Cereport and Carboplatin With Radiation Therapy for Children With Newly-Diagnosed Brain Stem Gliomas
Brief Title: Radiation Therapy Plus Carboplatin and Lobradimil in Treating Children With Newly Diagnosed Brain Stem Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ADVL0012; COG-ADVL0012 (Other: Children's Oncology Group); CCG-ADVL0012 (Other: Children's Cancer Group); ALK-01-042; CCG-09802 (Other: Children's Cancer Group); CDR0000067715 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Carboplatin; RMP 7; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Radiation Therapy, 33 Doses; Carboplatin 35mg^m2 for 20 Days (Experimental)
  Interventions: Drug: carboplatin; Drug: cereport; Radiation: radiation therapy
- Radiation Therapy, 33 Doses; Carboplatin 35mg^m2 for 25 Days (Experimental)
  Interventions: Drug: carboplatin; Drug: cereport; Radiation: radiation therapy
- Radiation Therapy, 33 Doses; Carboplatin 35mg^m2 for 30 Days (Experimental)
  Interventions: Drug: carboplatin; Drug: cereport; Radiation: radiation therapy
- Radiation Therapy, 33 Doses; Carboplatin 35mg^m2 for 33 Days (Experimental)
  Interventions: Drug: carboplatin; Drug: cereport; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
  Other Names: Paraplatin; CBDCA; NSC #241240
Drug: cereport
  Other Names: labradimil; IND #60315
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as carboplatin and lobradimil may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of combining radiation therapy with carboplatin and lobradimil in treating children who have newly diagnosed brain stem gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated duration of lobradimil plus carboplatin with radiotherapy in patients with newly diagnosed brain stem gliomas.
* Determine the toxic effects of this treatment regimen in these patients.
* Assess the response to radiotherapy in patients treated with this regimen.

OUTLINE: Patients receive radiotherapy for 5 consecutive days a week for 6.5 weeks, for a total of 33 doses. Patients receive carboplatin IV over 15 minutes followed by lobradimil IV over 10 minutes concurrently with radiotherapy.

The first cohort of 3-6 patients receives treatment with carboplatin and lobradimil for the first three weeks of radiotherapy, with the duration of chemotherapy increasing by one week with each subsequent cohort until the maximum duration of 6.5 weeks is reached or until unacceptable toxicity occurs in 2 of 6 patients.

Patients are followed at 6 weeks; every 3 months for 2 years; every 6 months for 3 years; and then annually thereafter.

PROJECTED ACCRUAL: A total of 15-24 patients will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed diffuse, intrinsic brain stem gliomas
* Measurable disease
* No disseminated disease at sites other than brain stem
* No neurofibromatosis
* Treatment must begin within 31 days of diagnosis

  * Date of diagnosis will be considered date of surgery in patients undergoing surgical biopsy

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Karnofsky 50-100% (over 10 years of age)
* Lansky 50-100% (10 years of age and under)

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGPT no greater than 2.5 times ULN (4.0 times ULN with antiepileptic or steroid medications)

Renal:

* Creatinine less than ULN for age OR
* Creatinine clearance or glomerular filtration rate greater than 80 mL/min

Other:

* No history of severe allergic reaction to any platinum-containing compound
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent growth factors during therapy with carboplatin

Chemotherapy

* Not specified

Endocrine therapy

* Prior corticosteroids for brain stem glioma are allowed

Radiotherapy

* Not specified

Surgery

* Prior surgery for brain stem glioma is allowed

Other

* At least 24 hours since any of the following medications:

  * Vasodilating compounds
  * Angiotensin-converting enzyme inhibitors
  * Calcium channel blockers
  * Beta blockers
* No other prior therapy for brain stem glioma

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2001-02; Primary Completion 2005-01 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival
  A MRI scan will be performed six (6) weeks after completion of radiation, plus at three-month intervals thereafter for two years, as long as there is no evidence of progressive disease. Children who are progression-free two years after treatment will have MRI scanning at six-month intervals, thereafter, for three more years

CONTACTS AND LOCATIONS:
Overall Officials: Roger J. Packer, MD, Study Chair — Children's National Research Institute
Locations (19):
- United States (19):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington